CLINICAL TRIAL: NCT06619717
Title: Optimizing Hyperbaric Oxygen Treatments for Acute Carbon Monoxide Poisoning: An Open-label Randomized Study.
Brief Title: Optimal Number of Hyperbaric Oxygen Treatments for Carbon Monoxide Poisoning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00146529
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Hyperbaric Oxygen Therapy; Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single HBO treatment (Active Comparator): The exact parameters of each dive will be left to individual clinicians. Commonly used treatments would be:
  1 treatment: 100% oxygen at 2.8 atmospheres for 30 minutes followed by a 10-minute air break, then 100% oxygen at 2 atmospheres for 60 minutes with one 10-minute air break after 30 minutes
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- Three HBO treatments (Experimental): The exact parameters of each dive will be left to individual clinicians. Commonly used treatments would be:
  3 treatments: Weaver protocol or similar variation (i.e. 100% oxygen at 3 atmospheres for 90 minutes with two 10-minute air breaks every 30 minutes. This will be repeated every 8 hours until 3 treatments are complete.)
  Interventions: Procedure: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — Three treatments with hyperbaric oxygen therapy. The exact parameters of each dive will be left to individual clinicians. Commonly used treatments would be:
  Weaver protocol, or similar (i.e. 100% oxygen at 3 atmospheres for 90 minutes with two 10-minute air breaks every 30 minutes. Repeat this every 8 hours until 3 treatments are complete.)
  Arms: Three HBO treatments
Procedure: Hyperbaric Oxygen Therapy — Single treatment with hyperbaric oxygen. Exact parameters left to treating physician but commonly: 100% oxygen at 2.8 atmospheres for 30 minutes followed by a 10-minute air break, then 100% oxygen at 2 atmospheres for 60 minutes with one 10-minute air break after 30 minutes
  Arms: Single HBO treatment

SUMMARY:
The optimal treatment strategy with hyperbaric oxygen therapy has been the subject of some debate over the past 3 decades. Initial landmark studies showed a decrease in the incidence of DNS with a single treatment and also with three treatments over the course of 24 hours. These two strategies have continued to be used widely without further evidence comparing them in a direct fashion. Retrospective publications in the years since have been largely conflicting about the benefit of additional hyperbaric treatments. The investigators would seek to randomize patients with carbon monoxide poisoning to receive with 1 or 3 treatments with hyperbaric oxygen and measure their neurologic outcomes.

DETAILED DESCRIPTION:
HBO is a niche treatment modality, especially in Canada. There are few sites which offer this care, and as such, treatment often carries significant logistical challenges. Since 2021, the HBO unit at the Misericordia hospital has averaged 49 patients per year being treated for CO poisoning. This HBO unit provides coverage to patients within Alberta, Saskatchewan, Manitoba, Yukon, and Northwest Territories. Due to the significant barriers to treatment, including the high cost to the public system, it is important to clearly understand how to best treat these patients.

Purpose:

The aim of this study is to assess whether a single treatment session of hyperbaric oxygen is non-inferior to three treatments for patients with acute carbon monoxide poisoning.

ELIGIBILITY:
Inclusion Criteria:

* All adult (over 17 years old) patients referred to a Hyperbaric Unit for acute carbon monoxide poisoning.

Exclusion Criteria:

* Obtunded
* Mechanically ventilated
* Pregnant
* Incarcerated
* Cognitively impaired (acutely or chronically)

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing delayed neurologic sequalae | 6 weeks and 6 months
  DNS includes a spectrum of symptoms such as depression, anxiety, memory issues, ataxia, behavioral changes, decreased cognitive function. For CO-poisoned patients who do not succumb to the direct effects of hypoxia, DNS is one of the primary causes of long-term morbidity.
  The presence of delayed neurologic sequelae as measured by a series of standardized tests. These tests will include digit span (Attention), the Boston Naming Test 15 (aphasia), general orientation and delayed recall (memory), and clock drawing (visuospatial). DNS will be considered present if a patient scores ≥2 SD below the standardized T scores for any neuropsychological test, if they score ≥1 SD below the standardized T scores for 2 or more tests, or if they score ≥1 SD below the standardized T score for any test and self-report poor memory/concentration/attention.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rowe, MD, MSc, CCFP (EM), FCCP, Study Director — Professor in the Department of Emergency Medicine, Faculty of Medicine & Dentistry, College of Health Sciences, at the University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No